CLINICAL TRIAL: NCT04865055
Title: Clinical Evaluation of the Photo-protective Efficacy of a Sunscreen (FLA No: 758637 10 and 758637 15) Product in Healthy Adults Volunteers for 7 Days
Brief Title: Photoprotection Efficacy With Sunscreen Formulas Containing the Cyclic Merocyanine Long-UVA Absorber MCE, Under Real Sun Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14CSI044
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Real Life Pigmentation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyclic merocyanine (Active Comparator): cyclic merocyanine long-UVA absorber
  Interventions: Other: cyclic merocyanine
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: cyclic merocyanine — long-UVA absorber
  Arms: cyclic merocyanine
Other: placebo — placebo
  Arms: placebo

SUMMARY:
To evaluate the photo-protector effect of BC_3 (E212657) formulated in SPF30 compared to SPF30 alone on real sun exposure induced pigmentation in healthy volunteers

DETAILED DESCRIPTION:
The study intends to evaluate the clinical efficacy of the photo-protective cosmetic products (758637 10 and 758637 15) and to compare the photo-protection potential of the two products, after its application for 7 days on healthy female volunteers under the normal conditions of use planned by the sponsor. The study will also evaluate the tolerance of the two products on the skin of healthy female volunteers.

The photo-protection is generally concerned with the reduction of exposure to ultra violet radiations, specifically UV-B and UV-A, primarily from the sun. The harmful radiations from the sun can cause various skin issues which can be as minor as skin tanning and as major as skin cancer. The photo-protective products can help in protection of the skin from the harmful sun radiation either by blocking them or absorbing them and preventing the rays to damage the skin

The formula number of both the products are 758637 10 and 758637 15. The SPF value of both the product is 30.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a healthy female volunteer aged between 18-45 years old
* Subjects with skin phototype IV-V and ITA° 4° to 20°.
* Subject who has given freely his or her informed consent and who is cooperative and aware of the necessity and duration of the controls so that perfect adherence to the protocol can be expected
* Subject who is able to read and understand documents transmitted (information sheet and consent form)
* If the subject is a female of childbearing potential and is willing to use a reliable mean of contraception*(for at least one month before the beginning of the study, and throughout the study) or menopausal women (absence of menstrual periods for one year or more)
* Accepting to stop the usage of all facial skin cosmetics (lotion, cream, powder, make-up) throughout the study duration.
* Subject willing to expose / her face and arms to sun for around 1- 2 hours morning and 1-2 hours afternoon during the day

  * sexually active females of childbearing potential should either be surgically sterile (oophorectomy, hysterectomy ortubal ligation), or should use a medically accepted contraceptive regimen: systemic contraceptive (oral, implant,injection), diaphragm or cervical cap, Intravaginal device, intrauterine device (IUD), condoms.

Exclusion Criteria:

* Female subject who is pregnant (as demonstrated by positive UPT on screening visit) or planning to get pregnant during the study.
* Female subjects who are breast-feeding.
* Subject with a known history or present condition of allergic response to any cosmetic products.
* Subject with photosensitive dermatosis (sensitive to sun exposure).
* Subject having skin diseases (e.g. moderate to severe acne vulgaris or nodulocystic acne, psoriasis,naevi, freckles, excess hair, uneven skin tones, vitiligo, active atopic dermatitis, pigmented contact dermatitis or other cutaneous manifestations),on face and upper portion of arms which can interfere with the test readings.
* Any treatment, topical or systemic, taken in the weeks preceding the screening, which is likely to interfere with the evaluation of the efficacy of the product(s) being studied.
* Subject undergoing anti-inflammatory, corticoids or retinoids therapy by oral or topical way
* Subject having used de-pigmenting products, masks exfoliant product on the investigational areas in last 4 weeks.
* Subject who has been deemed by the investigator as potentially unable or unwilling to comply with the protocol
* Subject enrolled in another clinical trial during the study period
* Personnel of the investigational site.
* Subject with any scar or tatoo on the investigational areas specifically on the face and upper arms

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-29 (Estimated); Primary Completion 2021-04-29 (Estimated); Study Completion 2021-04-29 (Estimated)

PRIMARY OUTCOMES:
To compare the photo-protective efficacy of two cosmetic investigational products by Clinical scoring done by the study investigator | Change from baseline at Day 7
  color chart
To compare the photo-protective efficacy of two cosmetic investigational products by Non invasive bio-instrumental skin color assessments | Change from baseline at Day 7
  Chromameter
To compare the photo-protective efficacy of two cosmetic investigational products by Self assessment | Change from baseline at Day 7
  questionnaire

SECONDARY OUTCOMES:
To evaluate the tolerance of both the photo protective cosmetic products (A - 758637 10 and B - 758637 15) | Change from baseline at Day 7
  The local intolerances reported by the subjects and observed by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- CIDP Biotech India Pvt. Lt, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: DECEMBER 2021